CLINICAL TRIAL: NCT04672226
Title: A Feasibility Study to Evaluate PDE MAX, a Food for Special Medical Purposes (FSMP) for Use in the Dietary Management of Pyridoxine Dependent Epilepsy (PDE) With Regards to Acceptability, Tolerability, Adherence and Effect on Metabolic Control
Brief Title: Evaluation of PDE MAX
Acronym: PDE MAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Collaborators: Radboud University Medical Center (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCT-W-PDEPS-2017-10-11; 254178 (Other: UK IRAS); 20/NW/0370 (Other: UK HRA)
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Pyridoxine Dependant Epilepsy
Keywords: PDE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDE MAX (Experimental): PDE MAX will be prescribed by the study dietitian based on the patient's individual requirement.
  Interventions: Dietary Supplement: PDE MAX

INTERVENTIONS:
Dietary Supplement: PDE MAX — PDE MAX will be prescribed by the study dietitian based on the patient's individual requirement.

SUMMARY:
PDE MAX is a single arm prospective, feasibility study in up to 15 participants aged one (1) year and over of PDE MAX for the dietary management of Pyridoxine Dependent Epilepsy.

DETAILED DESCRIPTION:
PDE Max is a newly-developed product designed specifically to meet the nutritional requirements of patients following a lysine-restricted diet for PDE.

This is a feasibility study to evaluate PDE MAX, a food for special medical purposes (FSMP) for use in the dietary management of Pyridoxine Dependent Epilepsy (PDE) with regards to acceptability, tolerability, adherence and effect on metabolic control.

Participants will be given an eight-week supply of PDE MAX and they will be asked to complete a daily diary and short questionnaire to record information on: adherence, gastrointestinal tolerance, palatability and how the product is used.

Blood and urine samples will be taken at the beginning and end of the study to measure several biochemical parameters.

Physical and neurological assessments will be carried out by the local Metabolic Consultant at the beginning and end of the study.

Routine monitoring of lysine levels will continue.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Pyridoxine Dependent Epilepsy (PDE), biochemically and/or genetically confirmed.
* Males or females aged one (1) year and above. Any participant aged 16 years and over at screening must have the capacity to consent for themselves.
* Currently following a lysine-restricted diet for a minimum of four (4) weeks prior to screening.
* Willing to take the study product and follow advice given by the dietitian.
* Willingly given, written, informed consent from patient or parent/guardian.
* Willingly given, written assent (if appropriate).

Exclusion Criteria:

* Inability to comply with the study protocol, in the opinion of the investigator.
* Use of additional macro/micronutrient supplements during the study period, unless clinically indicated and prescribed by the investigator, such as but not limited to arginine and pyridoxine. In which case, supplementation must have started four (4) weeks prior to screening with no anticipated changes to intakes during the study duration.
* Participants who are pregnant / breastfeeding at the start of the study or planning to become pregnant during the study period. Participants of child-bearing potential will be required to undergo pregnancy test prior to enrolment.

N.B.: Participants who become pregnant unexpectedly during this study may, in consultation with their doctor, continue on the study's dietary product if they wish but will not have any investigations that would not normally be carried out during pregnancy.

* Allergy to any ingredient present in the study product.
* Other concurrent medical or psychiatric conditions, which, in the opinion of the Investigator, would place the subject at increased risk, preclude obtaining voluntary consent/assent or compliance with required study procedures, or would confound the objectives of the study.
* Is participating in any other interventional study and has received any other investigational drug, product or device within 30 days prior to screening or are taking part in a non-medication study which, in the opinion of the investigator, would interfere with study compliance or outcome assessments.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Product acceptability rated on a Likert scale by the patient after eight week intake | 8 weeks
  Assessment of participant's acceptability following an eight week intake of the study product
Questionnaire of self-reported changes in gastrointestinal tolerance during eight week intake | 8 weeks
  Assessment of participant's gastrointestinal tolerance during the eight week intake of the study product
Questionnaire of self-reported adherence to the prescribed amount of study product | 8 weeks
  Assessment of participant's adherence to prescribed amount during the eight week intake of the study product

SECONDARY OUTCOMES:
Change in concentration from baseline, after an 8-week intake of PDE MAX, of pipecolic acid in plasma. | Day 0 (visit 1) to day 56 (visit 2)
  To observe any change from baseline, after an 8-week intake of PDE MAX, in pipecolic acid in plasma.
Change in concentration from baseline, after an 8-week intake of PDE MAX, of 6-oxo-pipecolic acid in bloodspots | Day 0 (visit 1) to day 56 (visit 2)
  To observe the changes from baseline, after an 8-week intake of PDE MAX, in 6-oxo-pipecolic acid in bloodspots
Change in concentration from baseline, after an 8-week intake of PDE MAX, of 6-oxo-pipecolic acid in plasma | Day 0 (visit 1) to day 56 (visit 2)
  To observe any changes from baseline, after an 8-week intake of PDE MAX, of 6-oxo-pipecolic acid in plasma
Change in concentration from baseline, after an 8-week intake of PDE MAX, of 6-oxo-pipecolic acid in urine | Day 0 (visit 1) to day 56 (visit 2)
  To observe any changes from baseline, after an 8-week intake of PDE MAX, of 6-oxo-pipecolic acid in urine
Change in concentration from baseline, after an 8-week intake of PDE MAX, of P6C in bloodspots | Day 0 (visit 1) to day 56 (visit 2)
  To observe any changes from baseline, after an 8-week intake of PDE MAX, of P6C in bloodspots
Change in concentration from baseline, after an 8-week intake of PDE MAX, of P6C in plasma | Day 0 (visit 1) to day 56 (visit 2)
  To observe any changes from baseline, after an 8-week intake of PDE MAX, of P6C in plasma
Change in concentration from baseline, after an 8-week intake of PDE MAX, of αAASA in plasma | Day 0 (visit 1) to day 56 (visit 2)
  To observe any changes from baseline, after an 8-week intake of PDE MAX, of αAASA in plasma
Change in concentration from baseline, after an 8-week intake of PDE MAX, of αAASA in urine | Day 0 (visit 1) to day 56 (visit 2)
  To observe any changes from baseline, after an 8-week intake of PDE MAX, of αAASA in urine
Change in concentration from baseline, after an 8-week intake of PDE MAX, of the amino acid profile in plasma | Day 0 (visit 1) to day 56 (visit 2)
  To observe any changes from baseline, after an 8-week intake of PDE MAX, of the amino acid profile in plasma
Change in concentration from baseline, after an 8-week intake of PDE MAX, of whole blood serotonin | Day 0 (visit 1) to day 56 (visit 2)
  To observe any changes from baseline, after an 8-week intake of PDE MAX, of whole blood serotonin
Change in concentration from baseline, after an 8-week intake of PDE MAX, of pyridoxal phosphate in plasma | Day 0 (visit 1) to day 56 (visit 2)
  To observe any changes from baseline, after an 8-week intake of PDE MAX, of pyridoxal phosphate in plasma
Change in concentration from baseline, after an 8-week intake of PDE MAX, of vitamers in plasma | Day 0 (visit 1) to day 56 (visit 2)
  To observe any changes from baseline, after an 8-week intake of PDE MAX, of vitamers in plasma
Change in concentration from baseline, after an 8-week intake of PDE MAX, of organic acids in urine | Day 0 (visit 1) to day 56 (visit 2)
  To observe any changes from baseline, after an 8-week intake of PDE MAX, of organic acids in urine
Change in concentration from baseline, after an 8-week intake of PDE MAX, of 2OPP in bloodspots | Day 0 (visit 1) to day 56 (visit 2)
  To observe the changes from baseline, after an 8-week intake of PDE MAX, of 2OPP in bloodspots
Change in concentration from baseline, after an 8-week intake of PDE MAX, of 2OPP in plasma | Day 0 (visit 1) to day 56 (visit 2)
  To observe the changes from baseline, after an 8-week intake of PDE MAX, of 2OPP in plasma
Change in concentration from baseline, after an 8-week intake of PDE MAX, of 2OPP in urine | Day 0 (visit 1) to day 56 (visit 2)
  To observe the changes from baseline, after an 8-week intake of PDE MAX, of 2OPP in urine

CONTACTS AND LOCATIONS:
Overall Officials: Clara van Karnebeek, Principal Investigator — Amsterdam University Medical Centers
Locations (2):
- Radboud UMC, Nijmegen, Netherlands
- Great Ormond Street Hospital for Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No